CLINICAL TRIAL: NCT05699174
Title: PO Versus IV Antibiotics for the Treatment of Infected Nonunion of Fractures After Fixation
Brief Title: PO vs IV Antibiotics for the Treatment of Infected Nonunion of Fractures After Fixation
Acronym: POvIV2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH2210635
Record Dates: First submitted 2023-01-11; First posted 2023-01-26 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-05

CONDITIONS: Infections; Infected Wound; Nonunion of Fracture; Injury Leg; Amputation; Internal Fixation; Complications, Infection or Inflammation; Fracture; Lower Extremity Fracture; Antibiotic Side Effect
MeSH Terms: conditions — Infections; Wound Infection; Fractures, Ununited; Leg Injuries; Inflammation; Fractures, Bone | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Two arm, randomized controlled multicenter Phase III trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care PO (oral) antibiotics (Active Comparator): An intervention in this study includes randomization of patients with an infected nonunion to standard of care PO (oral) antibiotics for up to 6 weeks post hospitalization. No medications will be provided by the study. Study participants will be prescribed their oral antibiotics by their treating physician and the specific type will depend on their infection diagnosis. Medications will be obtained using health insurance and/or resources available at the treating facility therefore the mode of antibiotics utilized as standard of care will vary across participating sites. Sites will follow their standard of care delivery for antibiotics and the study will defer to this standard.
  Interventions: Drug: Standard of Care PO (oral) antibiotics
- Standard of Care Intravenous (IV) antibiotics (Active Comparator): An intervention in this study includes randomization of patients with an infected nonunion to intravenous (IV) antibiotics for up to 6 weeks post hospitalization. No medications will be provided by the study. Study participants will be prescribed their IV antibiotics by their treating physician and the specific type will depend on their infection diagnosis. Medications will be obtained using health insurance and/or resources available at the treating facility therefore the mode of antibiotics utilized as standard of care will vary across participating sites. Sites will follow their standard of care delivery for antibiotics and the study will defer to this standard.
  Interventions: Drug: Standard of Care Intravenous (IV) antibiotics

INTERVENTIONS:
Drug: Standard of Care PO (oral) antibiotics — An intervention in this study includes randomization of patients with an infected nonunion to PO (oral) antibiotics for up to 6 weeks post hospitalization. The exact type of oral antibiotic will be depended on the patient's infection diagnosis.
  Arms: Standard of Care PO (oral) antibiotics
Drug: Standard of Care Intravenous (IV) antibiotics — An intervention in this study includes randomization of patients with an infected nonunion to intravenous (IV) antibiotics for up to 6 weeks post hospitalization. The exact type of IV antibiotic will be depended on the patient's infection diagnosis.
  Arms: Standard of Care Intravenous (IV) antibiotics

SUMMARY:
This is a Phase III clinical randomized control trial to investigate differences between patient with an infected nonunion treated by PO vs. IV antibiotics. The study population will be 250 patients, 18 years or older, being treated for infected nonunion after internal fixation of a fracture with a segmental defect less than one centimeter. Patients will be randomly assigned to either the treatment (group 1) PO antibiotics for 6 weeks or the control group (group 2) IV antibiotics for 6 weeks. The primary hypothesis is that the effectiveness of oral antibiotic therapy is equivalent to traditional intravenous antibiotic therapy for the treatment of infected nonunion after fracture internal fixation, when such therapy is combined with appropriate surgical management. Clinical effectiveness will be measured as the primary outcome as the number of secondary re-admissions related to injury and secondary outcomes of treatment failure (re-infection, nonunion, antibiotic complications) within the first one year of follow-up, as defined by specified criteria and determined by a blinded data assessment panel. In addition, treatment compliance, the cost of treatment, the number of surgeries required, the type and incidence of complications, and the duration of hospitalization will be measured.

DETAILED DESCRIPTION:
This is a Phase III clinical randomized control trial to investigate differences between patient with an infected nonunion treated by PO vs. IV antibiotics. The study population will be 250 patients, 18 years or older, being treated for infected nonunion after internal fixation of a fracture with a segmental defect less than one centimeter. Patients will be randomly assigned to either the treatment (group 1) PO antibiotics for 6 weeks or the control group (group 2) IV antibiotics for 6 weeks. The primary hypothesis is that the effectiveness of oral antibiotic therapy is equivalent to traditional intravenous antibiotic therapy for the treatment of infected nonunion after fracture internal fixation, when such therapy is combined with appropriate surgical management. Clinical effectiveness will be measured as the primary outcome as the number of secondary re-admissions related to injury and secondary outcomes of treatment failure (re-infection, nonunion, antibiotic complications) within the first one year of follow-up, as defined by specified criteria and determined by a blinded data assessment panel. In addition, treatment compliance, the cost of treatment, the number of surgeries required, the type and incidence of complications, and the duration of hospitalization will be measured.

The specific Aims of this study are to:

Specific Aim 1. Evaluate the effect of treatment of infected nonunion in bone fractures treated with revision fixation and either: (Group 1) operative debridement and PO antibiotic suppression for 6 weeks; or (Group 2) operative debridement and 6 weeks IV antibiotics.

Primary Hypothesis 1a: The rate of re-hospitalization for injury-related complication by one year in Group 1 will be non-inferior to the rate in Group 2.

Hypothesis 1b:. The rate of treatment failure by one year in Group 1 will be non-inferior to the rate in Group 2.

Hypothesis 1c: The rate of persistent infection by one year in Group 1 will be non-inferior to the rate in Group 2.

Hypothesis 1d: The rate of persistent nonunion by one year in Group 1 will be non-inferior to the rate in Group 2.

Hypothesis 1e: The rate of amputation by one year in Group 1 will be non-inferior to the rate in Group 2. Hypothesis 1f: Per patient total costs at 1 year will be lower in Group 1 than in Group 2.

Hypothesis 1g: Compliance in Group 1 will be non-inferior to compliance in Group 2.

Specific Aim 2. Build and validate a risk prediction model for failure of treatment of infected nonunion after fixation of fractures.

Hypothesis 2a: Demographic and injury characteristics will be highly predictive of treatment failure.

Hypothesis 2b: Open fractures will have a higher treatment failure rate than closed fractures.

Hypothesis 2c: Lower extremity fractures will have a higher treatment failure rate than upper extremity fractures.

Hypothesis 2d: Multiple organism infections will have a higher treatment failure rate than single organism infections.

Hypothesis 2e: Gram positive infections will have a higher treatment failure rate than gram negative infections.

Hypothesis 2f: Revision fixation with IMN and treatment failure will be non-inferior to the rate of treatment failure in revision fixation with plates.

Hypothesis 2g: Revision fixation with external fixation and treatment failure will be non-inferior to the rate of treatment failure in revision fixation with IMN or plates.

Hypothesis 2h: One Stage revision fixation strategies will be non-inferior to the rate of treatment failure in Two Staged revision fixation strategies

Study design: At time of treatment for infected nonunion, patients will be randomized to oral (PO) antibiotics group or intravenous (IV) antibiotics group. Patients will receive PO or IV antibiotics for 6 weeks at discharge from the hospitalization to treat the infected nonunion. Both groups will otherwise receive standard care treatment by attending orthopedic surgeon and healthcare team, including debridement and soft tissue coverage of wounds; laboratory evaluation of inflammatory markers at 2 weeks, and 6 weeks; clinical follow at 2 weeks, 6 weeks, 3 months, 6 months, and 12 months to assess recurrence of wound infection; and radiographic follow up at 6 weeks and 3 months or until boney union is confirmed.

Follow-Up: Assessments at baseline and at 2 weeks, 6 weeks, 3 months, 6 months and 12 months following hospital discharge will determine rates of re-hospitalization, treatment failure, infection, nonunion and amputation and patient compliance with antibiotic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Nonunion of a fracture that has previously undergone fixation. A Nonunion is defined as unplanned surgery with the primary purpose to promote union based on clinical/radiographic evidence >3 months after last fixation
2. Infection as determined by either

   1. FRI criteria
   2. CDC criteria (without the timeframe) This includes the possibility of culture negative, but determined to be infection by treating surgeon
3. Systemic antibiotic treatment regimen scheduled for at least 6 weeks

Exclusion Criteria:

1. Patients with a high risk of amputation based on the initial managing physician
2. Patients undergoing treatment of any other investigational therapy within the month preceding infection treatment or planned within the 12 months following infection treatment
3. Incarcerated or institutionalized patients
4. Patients who are unable to return for required follow-up visits and/or medical co-morbidities which preclude treatment with a general anesthetic
5. Patients with a prior history of chronic infection at the index site before fracture fixation
6. Patients with pathological fractures from a neoplastic process
7. History of Paget's Disease
8. The patient, or a designated proxy, unwilling to provide consent
9. The patient must be available for follow-up for at least 12 months following infection treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a hospital re-admission | 1 year
  Total number of re-admissions after revision fixation over the first 365 days post discharge from the hospitalization for initial surgical treatment of the infected nonunion. Re-admission can be for infection, nonunion, soft tissue revision, line complication, or antibiotic complication.

SECONDARY OUTCOMES:
Number of patients with treatment failure | 1 year
  Treatment Failure will define as patients with the following complications:
  * Wound problems requiring surgery
  * Patients that have culture positive recurrence of infection
  * Progressive radiographic loosening of the implant
  * Joint erosion due to infection
  * Infection with a new organism
  * Adverse reactions to any of the antibiotics
  * Infection recurrence
  * Persistent Nonunion
Number of patients with a re-hospitalization for a complication | 1 year
  Re-hospitalization for Complication is defined as:
  1. any re-admission to the hospital secondary to the treatment of the deep wound infection associated with the index fracture fixation for a defined set of complications. The list of complications includes: nonunion, amputation, infection, flap failure, , This definition has successfully been used by the core centers in previous published prospective studies and is consistent with the data used to generate the study power estimate.
  2. any complication of IV access requiring rehospitalization including, but not limited to line sepsis, DVT in same extremity as IV access, pneumothorax, or line change due to malfunction.
Number of patients with an additional infection | 1 year
  Infection will be assessed either as systemic inflammation or surgical site infection.
Number of patients that experienced amputation | 1 year
  Amputation is defined as surgical procedure to remove part of an extremity due to persistent infection or nonunion on proximal to site on affected extremity.
Medical Costs | 1 year
  Medical Costs for the index hospitalization and subsequent hospitalizations (within one year) will be derived using hospital bills and professional fee charges. Costs will be calculated from charges at the revenue center/cost department line level using cost-to-charge ratios (CCRs) computed from the Medicare Cost Reports (MCRs) specific to the hospital and fiscal year of the hospital stay. Of particular interest will be charges and costs associated with the surgical procedures for bone grafting (control and treatment), days hospitalized, and costs for subsequent admissions for complications.
Patient Reported Outcomes | 1 year
  Patient Report Outcomes Measurement Information System Computer Adaptive Test item banks, a product of the NIH Roadmap for Medical Research. CATs present an advantage over traditional measures in that they target only the most relevant items to each patient and can thus be used to obtain precise measurements with 4-6 items, making assessment across multiple domains feasible. CATs can also extend the ceiling and floor of individual domains, potentially enhancing responsiveness. At any visit if a CAT cannot be administered, respondents will instead complete the appropriate short forms associated with the CAT measure. In this study the following PROMIS domains will be used: Physical function, & Pain Inference in addition to PROMIS Global. Scores are measured on a T-score metric from 0-100 with 50 being the mean and standard deviation of 10 in the general U.S. population. Scores are categorized as: 0-30 severe, 31-40 moderate, 41-50 mild, and 51 and greater within normal limits.
Physical and Psychosocial Function Assessment | 1 year
  Physical and Psychosocial Function Assessment including measurements of symptoms, functioning, and healthcare-related quality of life will be assessed using the Patient-Reported Outcomes Measurement Information System PROMIS Global-10. The PROMIS Global-10 short form consists of 10 items that assess general domains of health and functioning including overall physical health, mental health, social health, pain, fatigue, and overall perceived quality of life. PROMIS Global-10 scoring allows each of the individual items to be examined separately to provide specific information about perceptions of physical function, pain, fatigue, emotional distress, social health and general perceptions of health. Scores are measured on a T-score metric from 0-100 with 50 being the mean and standard deviation of 10 in the general U.S. population. Scores are categorized as: 0-30 severe, 31-40 moderate, 41-50 mild, and 51 and greater within normal limits.
Adherence | 6 months
  Adherence will be measured by the Morisky Medication Adherence Scale (MMAS-8) which is an widely used 8-item expansion of the 4-item Morisky Medication Adherence Scale. The MMAS-8 an 8-item structured, self-report measure that assesses medication adherence. The questions 1-7 require a dichotomous reply and address the common reasons for missing medications. Question 8 is measured using a 5-point Likert scale and addresses difficulty of remembering to take medications. Scores are summed from 0-8 with a 6 or more being considered as adherent to the medications.
Compliance | 6 months
  Compliance will also be measured by percent of doses of medication taken. If less than 80% of doses of any antibiotic medication is taken then patient will be considered non-compliant. Compliance will be evaluated as a continuous variable.

CONTACTS AND LOCATIONS:
Overall Officials: William Obremskey, MD, Principal Investigator — Vanderbilt Medical Center; Renan Castillo, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (13):
- United States (13):
  - Indiana University, Indianapolis, Indiana
  - University of Maryland , MD Department of Orthopaedics, Baltimore, Maryland
  - Sinai Hospital Baltimore, Baltimore, Maryland
  - Hennepin Health, Minneapolis, Minnesota
  - Jamaica Hospital Medical Center, Queens, New York
  - Atrium Health, Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Okalahoma College of Medicine, Oklahoma City, Oklahoma
  - Penn State University M.S. Hershey Medical Center, Hershey, Pennsylvania
  - Vanderbilt Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Washington Harborview Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No